CLINICAL TRIAL: NCT03817671
Title: The Clinical Outcome of Ultra-low Oxygen Tension on Post Thawed Human Blastocyst
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Principal Investigator, Salma El Tanbouly, Senior Clinical Embryologist, Ganin Fertility Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GFCST11991
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Embryo Development
Keywords: Thawed blastocyst; ultra low oxygen tension; 2%O2; Degree of expansion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (5% O2) (Other): After thawing, embryos will be cultured in 25 μl drop of pre-equilibrated dishes of media covered with a layer of oil for 1.5 hours at 5.7% CO2, 5% O2, and 89.3% N2 till embryo transfer
  Interventions: Other: 5% O2
- Experimental arm (2%O2) (Experimental): After thawing, embryos will be cultured in 25 μl drop of pre-equilibrated dishes of media covered with a layer of oil for 1.5 hours at 5.7% CO2, 2% O2, and 92.3% N2 till embryo transfer
  Interventions: Other: 2% O2

INTERVENTIONS:
Other: 5% O2 — Culturing embryos in 5% O2 just after thawing and till embryo transfer
  Arms: Control arm (5% O2)
Other: 2% O2 — Culturing embryos in 2% O2 just after thawing and till embryo transfer
  Arms: Experimental arm (2%O2)

SUMMARY:
The clinical outcome of Ultra-low oxygen tension on post thawed human blastocyst

DETAILED DESCRIPTION:
In vitro, Embryo development depends on several factors as temperature, pH, and oxygen in the surrounding environment of the embryo. Impaired culture conditions are highly correlated with poor embryo development. Oxygen is a powerful regulator of embryo function , as it is responsible for cell respiration, energy production and rapid cell growth . Increased levels of oxygen is associated with an increase in the levels of ROS , which leads to unfavorable culture conditions, as it might affect the stability of cell membrane, DNA, and protein function .

In the female reproductive tract, oxygen concentration fluctuates between 2-8%, which is considered to be at its highest level in the fallopian tube, while the lowest level is in the uterus . Pre-implantation embryo crosses the uterotubal junction after the time of compaction on Day 3, where it is exposed to a shift in oxygen tension to 2%. This variation may have a role in the metabolic reactions of the embryo, and in its preparation for implantation process.

Some studies suggested that culturing embryos with oxygen tension below 5% may have an embryological advantage mimicking nature.

Embryological laboratories routinely use low Oxygen tension (5%). Our purpose is to investigate if ultra-low oxygen tension (2%) has an advantage over low oxygen tension (5%) for post thawed human embryo regarding clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Single or Multiple Embryo transfer embryo transfer. Female age 18-40. Embryo vitrified on day 5 or day 6 of insemination.

Exclusion Criteria:

Use of sperm donation. Use of Oocyte donation. Use of gestational carrier. Uterine congenital anomalies. Presence of any of the endometrial factors that affect embryo implantation such as hydrosalpings, adenomyosis or previously known uterine infection.

Any contradictions to undergoing in vitro fertilization or gonadotropin stimulation.

Ages: 5 Days to 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy rate | Time frame: 15 days following embryo transfer
  Defined as the pregnancy that is confirmed by both high levels of hCG and ultrasound confirmation of a gestational sac or heartbeat

SECONDARY OUTCOMES:
Ongoing pregnancy rate | Time frame: 20 weeks of gestation
  Defined as the proportion of pregnancies that had completed ≥20 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Hosam Zaki, MSc, FRCOG, Study Chair — Ganin Fertility Center, Cairo, Egypt.; Salma El Tanbouly, BSc., Principal Investigator — Ganin Fertility Center, Cairo, Egypt.; Abd El Ghafar Hussin, BSc., Principal Investigator — Ganin Fertility Center, Cairo, Egypt.; Hanaa El Khedr, Principal Investigator — Ganin Fertility Center, Cairo, Egypt.
Locations (1):
- Ganin Fertility Center, Cairo, Egypt

REFERENCES:
- [Background] Swain JE, Carrell D, Cobo A, Meseguer M, Rubio C, Smith GD. Optimizing the culture environment and embryo manipulation to help maintain embryo developmental potential. Fertil Steril. 2016 Mar;105(3):571-587. doi: 10.1016/j.fertnstert.2016.01.035. Epub 2016 Feb 3. PMID 26851765
- [Background] Gardner DK. The impact of physiological oxygen during culture, and vitrification for cryopreservation, on the outcome of extended culture in human IVF. Reprod Biomed Online. 2016 Feb;32(2):137-41. doi: 10.1016/j.rbmo.2015.11.008. Epub 2015 Nov 25. PMID 26687905
- [Background] Morin SJ. Oxygen tension in embryo culture: does a shift to 2% O2 in extended culture represent the most physiologic system? J Assist Reprod Genet. 2017 Mar;34(3):309-314. doi: 10.1007/s10815-017-0880-z. Epub 2017 Feb 8. PMID 28181051
- [Background] Oliveira JB. Does embryo culture at low oxygen tension improve ART outcomes? JBRA Assist Reprod. 2017 Feb 1;21(1):1. doi: 10.5935/1518-0557.20170001. No abstract available. PMID 28333022
- [Background] Kaser DJ, Bogale B, Sarda V, Farland LV, Williams PL, Racowsky C. Randomized controlled trial of low (5%) versus ultralow (2%) oxygen for extended culture using bipronucleate and tripronucleate human preimplantation embryos. Fertil Steril. 2018 Jun;109(6):1030-1037.e2. doi: 10.1016/j.fertnstert.2018.02.119. PMID 29935641
- [Background] Ng KYB, Mingels R, Morgan H, Macklon N, Cheong Y. In vivo oxygen, temperature and pH dynamics in the female reproductive tract and their importance in human conception: a systematic review. Hum Reprod Update. 2018 Jan 1;24(1):15-34. doi: 10.1093/humupd/dmx028. PMID 29077897
- [Background] Yang Y, Xu Y, Ding C, Khoudja RY, Lin M, Awonuga AO, Dai J, Puscheck EE, Rappolee DA, Zhou C. Comparison of 2, 5, and 20 % O2 on the development of post-thaw human embryos. J Assist Reprod Genet. 2016 Jul;33(7):919-27. doi: 10.1007/s10815-016-0693-5. Epub 2016 Mar 23. PMID 27007876
- [Background] Leese HJ. Human embryo culture: back to nature. J Assist Reprod Genet. 1998 Sep;15(8):466-8. doi: 10.1023/a:1022526219202. No abstract available. PMID 9785193